CLINICAL TRIAL: NCT00525655
Title: Multimedia Intervention in Patients With Familial Adenomatous Polyposis (FAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006-1037; NCI-2011-02827 (Registry Identifier: NCI CTRP); 1R41CA126453-01A1 (NIH)
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Familial Adenomatous Polyposis; Colorectal Cancer
Keywords: Familial Adenomatous Polyposis; Colorectal Cancer; Multimedia Intervention; Questionnaire; Survey; FAP
MeSH Terms: conditions — Adenomatous Polyposis Coli; Colorectal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimedia Intervention (Experimental)
  Interventions: Behavioral: Web-Based Multimedia Intervention; Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Web-Based Multimedia Intervention — Website designed to offer information and support for adolescents and young adults with FAP, viewed for 30-60 minutes.
Behavioral: Questionnaire — Questionnaires taking 10-15 minutes to complete.
  Other Names: Survey

SUMMARY:
The goal of this research study is to test the first version of a website that will offer information and support for adolescents and young adults with FAP. Researchers want to see if the website will be helpful, easy to understand, and easy to use for young patients with FAP.

DETAILED DESCRIPTION:
Study Participation:

If you agree to take part in this study, you will view the website, take part in a one-on-one interview or a small group discussion (a focus group), and one or more questionnaires. You may come to M. D. Anderson to take part in this study, which may take place during your routine doctor visit, if this is possible. If you are enrolled in a registry outside of M. D. Anderson, or if you do not wish to come to M. D. Anderson, you will access the website over the internet.

You will be asked to fill out a brief knowledge and quality of life questionnaire that will take 10-15 minutes to complete. For the website, you will be asked to view (all or parts) of an early version. The website is designed to offer information and support for adolescents and young adults with FAP. Viewing the website will take about 30-60 minutes, depending on what stage of development the website is in at the time.

For the one-on-one interview or focus group (after viewing the website), you will speak with a research assistant. You will be asked for your permission to record this interview or focus group on an audiotape so that study staff can collect all of your responses. During this interview or focus group, you will be asked about different aspects of the website, including if you like it, if the information is useful to you, and if the website is easy to understand and use. You will also be asked about ways that you think the website can be improved or changed to better serve adolescents and young adults patients with FAP. This interview or focus group will take about 15-30 minutes to complete.

For the questionnaire, some participants (those who view later versions of the website) will also be asked to complete the Website Analysis and Measurement Inventory (WAMMI). The WAMMI is a questionnaire that will measure if the website is appealing and easy to use for adolescents and young adults patients with FAP. Examples of questions on the WAMMI will be about whether you can quickly find what you want on the website and whether everything on this website easy to understand. You will be able to answer the questions on a 5-point scale from "Strongly Agree" to "Strongly Disagree." The questionnaire will take about 5-10 minutes to complete.

After you have finished viewing the website and completed the interview (and/or questionnaire), you will be given the option to speak with a genetic counselor if you have any questions about FAP.

Length of Study:

Your total time on this study will range from about 45 minutes to 2 hours. Your participation will be over in this study once you have finished viewing the website and completed the interview and/or questionnaire.

This is an investigational study. Up to 55 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Eligibility: (List All Criteria)

Inclusion Criteria:

1. 1) Having a confirmed genetic or clinical diagnosis of FAP between the age of 13-24 at the time of recruitment to this study.
2. 18-21 year old with a previous cancer diagnosis.
3. Able to read and speak English.

Exclusion Criteria:

1) n/a

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Pilot Test FAP Website (Interviews) | 2 years

SECONDARY OUTCOMES:
Participant Assessment of FAP Website (Questionnaire) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Peterson, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org